CLINICAL TRIAL: NCT07009275
Title: Development of Game-based Simulation Application With 3D Animation Technology for Vital Signs Measurement Skills in Nursing Education
Brief Title: Game-Based 3D Simulation for Vital Signs Training in Nursing Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Collaborators: Sakarya University of Applied Sciences (Unknown)
Responsible Party: Principal Investigator, Funda Erol, Dr., Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: E-26428519-044-65435
Record Dates: First submitted 2025-05-20; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Nursing Education; Vital Signs; Animation; Academic Acheivement; Satisfaction
Keywords: nursing education; vital signs; animation; academic acheivement; satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: A randomized controlled experimental design
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group consisted of students using the game-based simulation application developed using 3D animation technology.
  Interventions: Other: The game-based simulation application developed using 3D animation technology
- Control group (No Intervention)

INTERVENTIONS:
Other: The game-based simulation application developed using 3D animation technology — The intervention group consisted of students using the game-based simulation application developed using 3D animation technology, while the control group consisted of students using traditional learning methods.
  Arms: Intervention group

SUMMARY:
This study aims to improve nursing students' skills in measuring vital signs using a 3D animation-based game simulation. Measuring vital signs is a key responsibility for nurses and requires both knowledge and hands-on practice. To help students learn without risking patient safety, we developed an educational game that uses 3D animation technology.

A total of 73 nursing students participated in this randomized controlled study. One group used the 3D game simulation, while the other group received traditional teaching. We compared students' test scores, their satisfaction with the learning method, and their confidence in what they learned.

DETAILED DESCRIPTION:
The nursing profession is a discipline that requires competence in both cognitive and psychomotor skills in order to protect and improve the health of individuals and provide appropriate care in cases of illness [1]. In this context, the effective acquisition of psychomotor skills is considered to be one of the fundamental objectives of nursing education [2]. During the education process, students are expected to acquire many skills of varying degrees of difficulty and complexity and become proficient in their application [3]. Among these skills, the accurate assessment, measurement and monitoring of vital signs is one of the important responsibilities of nurses [4].

Any change in vital signs is an early indicator of changes in the patient's overall condition [5, 6]. Therefore, accurate and timely monitoring of vital signs and their effective use in the clinical decision-making process are of great importance for patient safety [7]. However, the relevant literature indicates that vital signs are not regularly and accurately monitored by nurses, and that the quality of monitoring is poor or not reported [8, 9]. So, these omissions in monitoring vital signs lead to an increase in preventable intensive care admissions and mortality rates [10].

Monitoring vital signs, which is critical for effective patient management in clinics, is often left to nursing students with basic knowledge [11]. However, due to the non-invasive nature of vital signs applications, students often perform these applications with minimal or no supervision from a clinical nurse educators or nurses [12]. A review of the literature reveals significant deficiencies in students' knowledge and application of vital signs [11-13]. It is critical that students perform the clinical skills they have acquired correctly and appropriately in order to improve patient safety and quality of care [14, 15]. Considering the importance of monitoring vital signs in a timely and accurate manner for the early identification of clinical deterioration, nursing students must be competent in vital signs assessment [12]. Therefore, it is necessary to use more effective and current learning methods in teaching vital signs.

At this point, the integration of innovative technologies into nursing education enables students to gain experience by repeating these applications without harming the patient and learning from their mistakes [16]. One of these technologies is a virtual game simulation obtained by transferring a real-life situation to the computer platform and gamifying it, which has just begun to be used in nursing education [15]. Recently, virtual gaming simulations have been increasingly used in nursing education to reduce some of the resource challenges of face-to-face simulation [17]. The objective of a virtual gaming simulation is to provide students with the opportunity to apply the concepts they have learned in a realistic scenario [18]. This practice enables students to actively participate in their own learning by its very nature [19]. The utilisation of virtual gaming simulations affords students the opportunity to receive prompt feedback, oversee their performance and conduct objective assessments [20]. Students are afforded the opportunity to repeat the game until they are satisfied with their performance [21]. Therefore, virtual game simulations contribute to the increase of students' academic achievement and skill performance [20]. At the same time, virtual gaming simulation as a teaching strategy enables students to participate in a realistic clinical scenario, reducing their anxiety and supporting their self-confidence [15, 22]. Because simulation offers students the opportunity to develop their nursing knowledge, clinical and psychomotor skills and clinical decision making levels in a simulated safe environment and over a long period of time before encountering real patients [17].

When reviewing the literature on nursing education, no research findings were found regarding the use of game-based virtual reality simulation applications for measurement skills related to vital signs. In this study, a game-based simulation application developed using 3D animation technology was designed to fill this gap and to enable nursing students to acquire vital signs measurement skills. We aimed to evaluate the effects of this application on students' academic achievement, satisfaction and self-confidence in learning. In this way, the aim is to provide an effective and technology-based teaching strategy that will increase patient safety in nursing education.

ELIGIBILITY:
Inclusion Criteria:

* Being enrolled as a student in the Faculty of Nursing,
* Voluntarily agreeing to participate in the study,
* Not having previously received theoretical and practical training on vital signs,
* Not being an international student,
* Not having transferred to the Faculty of Nursing from other health sciences programs with different educational or assessment practices.

Exclusion Criteria:

* Not being enrolled in the Faculty of Nursing,
* Refusing to participate or withdrawing consent,
* Having prior theoretical or practical education related to vital signs,
* Being an international student,
* Having transferred from other health sciences programs that use different clinical or educational evaluation systems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
Academic Achievement Test of Vital Sings Measurement Skills | From enrollment to the end of implementation at 4 weeks
  The researchers developed the Academic Achievement Test of Vital Signs Measurement Skills to measure vital signs. The researchers first identified the gains that students should make in measuring vital signs. In line with the literature [6, 12, 13], five-choice multiple-choice questions were prepared covering the goals and behaviours determined for each outcome. A total of 58 questions, including 23 questions on blood pressure measurement skills, 12 questions on apical pressure measurement skills, 10 questions on body temperature measurement skills, 7 questions on pulse taking skills, and 6 questions on respiration counting skills, were submitted for expert opinion by email. The questions were rearranged according to the experts' feedback. The questions were administered to 303 nursing students and a pretest was conducted. Question items were analysed and validity and reliability analyses of the questions were performed. In the final stage, inappropriate questions were removed.

SECONDARY OUTCOMES:
Student Satisfaction and Self-Confidence in Learning Scale | From enrollment to the end of implementation at 4 weeks.
  The original scale was developed by Jeffries and Rizzolo (2006) as 13 items, and the total number of items was reduced to 12 during its adaptation to Turkish. The scale is 5-point Likert type and consists of the sub-items 'satisfaction with current learning' and 'confidence in learning'. Satisfaction with current learning sub-item consists of 5 items, confidence in learning sub-item consists of 7 items, and there are no negative items. The Cronbach alpha value of the scale is 0.85 for 'satisfaction with current learning', 0.77 for 'confidence in learning' and 0.89 for the total scale. As the total score obtained from the scale increases, so does the student's satisfaction and confidence in learning.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, İzmit, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yılmaz D, Çınar G. The effect of simulator use in blood pressure measurement training on nursing students' psychomotor skills. Sağlık ve Toplum Dergisi. 2020;20(1):104-10
- [Background] Bayram SB, Caliskan N. The use of virtual reality simulations in nursing education, and patient safety. Contemporary Topics in Patient Safety-Volume 1: IntechOpen; 2020
- [Background] Luctkar-Flude M, Tyerman J, Tregunno D, Bell C, Lalonde M, McParland T, et al. Designing a virtual simulation game as presimulation preparation for a respiratory distress simulation for senior nursing students: Usability, feasibility, and perceived impact on learning. Clinical Simulation in Nursing. 2021;52:35-42
- [Background] Bayram ŞB, Çalışkan N. Using a game-based virtual reality application in psychomotor skills acquisition: An experience sharing Journal of Human Sciences. 2019;16(1):155-63
- [Background] Verkuyl M, Hughes M. Virtual gaming simulation in nursing education: A mixed-methods study. Clinical Simulation in Nursing. 2019;29:9-14
- [Background] Atthill S, Witmer D, Luctkar-Flude M, Tyerman J. Exploring the impact of a virtual asynchronous debriefing method after a virtual simulation game to support clinical decision-making. Clinical Simulation in Nursing. 2021;50:10-8
- [Background] Şahin G, Başak T. Game-based learning in nursing education. Gümüşhane University Journal of Health Sciences. 2019;8(3):308-14
- [Background] Mohammed QH. Knowledge and practices of nursing college student's regarding blood pressure measurement in Hospitals at Kirkuk City. Kufa Journal for Nursing Sciences. 2016;6(2):177-84
- [Background] Özsaban A, Turan N, Beki Ç, Aşti T. The relationship between nurses' attitudes toward vital signs monitoring and emotional ıntelligence levels. Genel Tıp Dergisi. 2022;32(6):652-7
- [Background] Kısacık ÖG, Gündoğan AÖ, Yılmaz E. Attitudes of Nurses and Nursing Students Towards Vital Signs: A Comparatıve Study. Journal of Nursing Effect. 2024;17(4):575-90
- [Background] Gülnar E, Yılmaz ED, Özveren H. Hemşirelerin yaşam bulgularina ilişkin tutum ve uygulamalarinin belirlenmesi. Kırıkkale Üniversitesi Tıp Fakültesi Dergisi. 2020;22(3):377-85
- [Background] Öztürk D, Göçmen Baykara Z. The effect of peer education on the teaching of nursing skills. Journal of Education and Research in Nursing. 2019;16(4):295-300
- [Background] Foronda CL, Fernandez-Burgos M, Nadeau C, Kelley CN, Henry MN. Virtual Simulation in Nursing Education: A Systematic Review Spanning 1996 to 2018. Simul Healthc. 2020 Feb;15(1):46-54. doi: 10.1097/SIH.0000000000000411. PMID 32028447
- [Background] Ordu Y, Caliskan N. The effect of virtual game simulation on students' perception of nursing diagnosis and clinical practice: Post-test only randomized controlled trial. Nurse Educ Pract. 2023 Oct;72:103792. doi: 10.1016/j.nepr.2023.103792. Epub 2023 Sep 26. PMID 37769493
- [Background] Carrero-Planells A, Pol-Castaneda S, Alamillos-Guardiola MC, Prieto-Alomar A, Tomas-Sanchez M, Moreno-Mulet C. Students and teachers' satisfaction and perspectives on high-fidelity simulation for learning fundamental nursing procedures: A mixed-method study. Nurse Educ Today. 2021 Sep;104:104981. doi: 10.1016/j.nedt.2021.104981. Epub 2021 May 25. PMID 34062333
- [Background] Alshehry AS, Cruz JP, Bashtawi MA, Almutairi KO, Tumala RB. Nursing Students' Knowledge, Competence and Attitudes towards Vital Signs Monitoring during Clinical Practice. J Clin Nurs. 2021 Mar;30(5-6):664-675. doi: 10.1111/jocn.15586. Epub 2020 Dec 16. PMID 33259648
- [Background] Connor N, McArthur D, Camargo Plazas P. Reflections on vital sign measurement in nursing practice. Nurs Philos. 2021 Jan;22(1):e12326. doi: 10.1111/nup.12326. Epub 2020 Oct 1. PMID 33001547
- [Background] Gillan PC, Delaney LJ, Tutticci N, Johnston S. Factors influencing nursing students' ability to recognise and respond to simulated patient deterioration: A scoping review. Nurse Educ Pract. 2022 Jul;62:103350. doi: 10.1016/j.nepr.2022.103350. Epub 2022 Apr 20. PMID 35468343
- [Background] Kellett J, Sebat F. Make vital signs great again - A call for action. Eur J Intern Med. 2017 Nov;45:13-19. doi: 10.1016/j.ejim.2017.09.018. Epub 2017 Sep 20. PMID 28941841
- [Background] Mok W, Wang W, Cooper S, Ang EN, Liaw SY. Attitudes towards vital signs monitoring in the detection of clinical deterioration: scale development and survey of ward nurses. Int J Qual Health Care. 2015 Jun;27(3):207-13. doi: 10.1093/intqhc/mzv019. Epub 2015 Apr 16. PMID 25888564
- [Background] Kamio T, Kajiwara A, Iizuka Y, Shiotsuka J, Sanui M. Frequency of vital sign measurement among intubated patients in the general ward and nurses' attitudes toward vital sign measurement. J Multidiscip Healthc. 2018 Oct 15;11:575-581. doi: 10.2147/JMDH.S179033. eCollection 2018. PMID 30410344
- [Background] Eyikara E, Baykara ZG. Effect of simulation on the ability of first year nursing students to learn vital signs. Nurse Educ Today. 2018 Jan;60:101-106. doi: 10.1016/j.nedt.2017.09.023. Epub 2017 Oct 13. PMID 29078202
- [Derived] Tanrikulu F, Gundogdu H, Erol F, Dikmen Y. A comparison of 3D game-based simulation versus traditional methods in vital signs education. BMC Med Educ. 2025 Oct 2;25(1):1344. doi: 10.1186/s12909-025-07980-4. PMID 41039559